CLINICAL TRIAL: NCT01286012
Title: Physiological Iron Maintenance in End Stage Renal Disease (ESRD) Subjects by Delivery of Soluble Ferric Pyrophosphate (SFP) Via Hemodialysate: The PRIME Study
Brief Title: Continuous Soluble Ferric Pyrophosphate (SFP) Iron Delivery Via Dialysate in Hemodialysis Patients
Acronym: PRIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIH-FP-01 PRIME
Record Dates: First submitted 2011-01-18; First posted 2011-01-31 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-08

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease, Hemodialysis, SFP
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — spleen fibrinolytic proteinase (human); Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SFP in liquid bicarbonate (Active Comparator)
  Interventions: Drug: Soluble Ferric Pyrophosphate in liquid bicarbonate; Drug: Erythrocyte Stimulating Agent (ESA); Drug: Intravenous (IV) Iron
- Placebo: Conventional Liquid Bicarbonate (Placebo Comparator): Control concentrate lacking SFP does not contain SFP (total iron = 0)
  Interventions: Drug: Placebo: Conventional liquid bicarbonate; Drug: Erythrocyte Stimulating Agent (ESA); Drug: Intravenous (IV) Iron

INTERVENTIONS:
Drug: Soluble Ferric Pyrophosphate in liquid bicarbonate — Subjects will receive hemodialysis containing SFP at 2 µM (11 µg iron/dL of dialysate) at every dialysis session, for a total duration of 36 weeks.
  Other Names: SFP
  Arms: SFP in liquid bicarbonate
Drug: Placebo: Conventional liquid bicarbonate — Subjects will receive hemodialysis containing conventional liquid bicarbonate lacking SFP at every dialysis session, for a total duration of 36 weeks.
  Arms: Placebo: Conventional Liquid Bicarbonate
Drug: Erythrocyte Stimulating Agent (ESA) — ESA was administered according to the recommendation of a blinded central anemia management center (CAMC) based on the weekly hemoglobin value and its rate of change.
Drug: Intravenous (IV) Iron — Approved IV iron preparations were administered per a protocol driven algorithm when patients serum ferritin value decreased below 200 ug/L.

SUMMARY:
The purpose of this study is to compare the clinical safety and efficacy of SFP in sparing the need for erythropoiesis stimulating agents (ESAs) required to maintain hemoglobin (hgb) levels in chronic hemodialysis subjects who receive SFP via the dialysate versus subjects who receive conventional dialysate without iron.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male and female subjects ≥ 18 years of age.
2. End-stage renal disease undergoing maintenance hemodialysis 3 to 4 times a week for at least 4 months and expected to remain on this schedule and be able to complete the study. Subjects on a cadaveric transplant list need not be excluded for this reason unless there is an identified donor.
3. Mean Hgb in the range of ≥ 9.5 to ≤ 12.0 g/dL during screening.
4. The difference between the maximum and minimum Hgb values during screening does not exceed 1.0 g/dL.
5. Mean ferritin ≥ 200 to ≤ 1000 µg/L during screening.
6. Mean TSAT ≥ 15% to ≤ 40% during screening.
7. Any and all serum albumin measured during the 2 months preceding randomization must be ≥ 3.0 g/dL.
8. Prescribed ESA dosing remaining in the range of ≥ 4,000 to ≤ 45,000 U/week epoetin or ≥ 12.5 to ≤ 200 µg/week darbepoetin during the 6 weeks preceding randomization.
9. Required IV iron at any time in the 6 months preceding randomization.

Main Exclusion Criteria:

1. Vascular access for dialysis is a catheter.
2. During the 6 months prior to randomization, infection of the vascular access to be used at the time of randomization.
3. Received a total of > 600 mg IV iron during the 6 weeks prior to randomization.
4. Received any amount of IV or oral iron during the 2 weeks prior to randomization.
5. Change in prescribed ESA dose:

   1. Any change in prescribed ESA dose within 4 weeks prior to randomization.
   2. The prescribed ESA dose at the time of randomization is > 25% higher or lower than the prescribed dose at 6 weeks prior to randomization.
   3. Change in prescribed type of ESA (e.g., epoetin vs. darbepoetin) or route of administration within 6 weeks prior to randomization.
6. Actual ESA dosing missed or withheld for a cumulative total of ≥ 1 week for any reason during the 6 weeks prior to randomization.
7. Known cause of anemia other than anemia attributable to renal disease (e.g., sickle cell disease, thalassemia, pure red cell aplasia, hemolytic anemia, myelodysplastic syndrome, etc.)
8. Scheduled kidney transplant or a donor has been identified but the transplant has not been scheduled.
9. Known ongoing inflammatory disorder (other than Chronic Kidney Disease), such as systemic lupus erythematosus, rheumatoid arthritis, other collagen-vascular diseases, etc.

11. Known active tuberculosis, fungal, viral, or parasitic infection requiring anti-microbial therapy or anticipated to require anti-microbial therapy during the patient's participation in this study. Subjects with hepatitis C, in the absence of cirrhosis, are not excluded from participation in the study if Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels are below 2 times the upper limit of normal on a consistent basis during the 2 months preceding randomization.

12. Occult tuberculosis requiring prophylactic treatment with anti-tubercular drug(s) that overlaps with the patient's participation in this study.

13. Cirrhosis of the liver based on histological criteria or clinical criteria (e.g., presence of ascites, esophageal varices, spider nevi, or history of hepatic encephalopathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Pratt, MD, Study Director — Rockwell Medical
Locations (21):
- United States (20):
  - Investigator, Birmingham, Alabama
  - Investigator, Tempe, Arizona
  - Investigator, Granada Hills, California
  - Investigator, Colorado Springs, Colorado
  - Investigator, Miami, Florida
  - Investigator, Albany, Georgia
  - Investigator, Hayden, Idaho
  - Investigator, Louisville, Kentucky
  - Investigator, New Orleans, Louisiana
  - Investigator, Columbus, Mississippi
  - Investigator, Kansas City, Missouri
  - Investigator, Las Vegas, Nevada
  - Investigator, Paterson, New Jersey
  - Investigator, Lexington, North Carolina
  - Investigator, Columbia, Tennessee
  - Investigator, Duncanville, Texas
  - Investigator, Greenville, Texas
  - Investigator, San Antonio, Texas
  - Investigator, St. George, Utah
  - Investigator, Taylorsville, Utah
- Investigator, Fajardo, Puerto Rico

REFERENCES:
- [Derived] Gupta A, Lin V, Guss C, Pratt R, Ikizler TA, Besarab A. Ferric pyrophosphate citrate administered via dialysate reduces erythropoiesis-stimulating agent use and maintains hemoglobin in hemodialysis patients. Kidney Int. 2015 Nov;88(5):1187-94. doi: 10.1038/ki.2015.203. Epub 2015 Jul 8. PMID 26154926

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Conventional Liquid Bicarbonate: Control concentrate lacking SFP does not contain SFP (total iron = 0)
  Subjects will receive hemodialysis containing conventional liquid bicarbonate lacking iron (placebo) at every dialysis session, for a total duration of 36 weeks.
Period: Overall Study
Arm/Group | SFP in Liquid Bicarbonate | Placebo: Conventional Liquid Bicarbonate
Started | 54 (2 patients randomized to SFP did not receive study drug.) | 54 (3 patients randomized to placebo did not receive study drug.)
Completed | 41 | 40
Not Completed | 13 | 14
Not completed — Adverse Event | 3 | 3
Not completed — Death | 2 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Physician Decision | 2 | 0
Not completed — peritoneal dialysis, randomized in error | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety Population: Subjects who received any amount of study drug, including those who receive the wrong treatment.
Groups:
- SFP in Liquid Bicarbonate: Soluble Ferric Pyrophosphate in liquid bicarbonate: Subjects will be randomized in a 1:1 ratio to receive hemodialysis containing SFP at 2 µM (11 µg iron/dL of dialysate) or conventional solutions lacking iron (placebo) at every dialysis session, for a total duration of 36 weeks.
- Total: Total of all reporting groups
Arm/Group | SFP in Liquid Bicarbonate | Placebo: Conventional Liquid Bicarbonate | Total
Number analyzed (Participants) | 54 | 49 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (12.40) | 58.5 (13.89) | 59 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 31 | 32 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 17 | 39
  White | 31 | 32 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 21 | 41
  Not Hispanic or Latino | 34 | 28 | 62
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percent Change From Baseline in ESA Dose Required to Maintain Hemoglobin in the Target Range, Adjusted for Hgb.
Description: The statistical endpoint is the change from baseline between groups at End of Treatment, where the baseline prescribed ESA dose (expressed as U/week epoetin) per subject is defined as the average weekly dose of ESA prescribed for administration over the two-week period of time immediately prior to randomization. The end-of-treatment prescribed ESA dose (expressed as U/week epoetin) per subject is defined as the average weekly dose of ESA prescribed for administration over the last two weeks of the treatment period.
Time Frame: Hemoglobin measured weekly and serum ferritin and Transferrin Saturation (TSAT) determined every other week; ESA dose recorded at each visit for 36 weeks.
Population: MITT population: Randomized subjects who received at least one dose of study drug and also received ESA during the treatment period.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | SFP in Liquid Bicarbonate | Placebo: Conventional Liquid Bicarbonate
Number analyzed (Participants) | 52 | 51
Percent change | 4.9 (12.07) | 39.8 (12.18)
Statistical Analysis 1: Comparison: SFP in Liquid Bicarbonate vs Placebo: Conventional Liquid Bicarbonate; Test type: Superiority or Other; p < 0.05, ANCOVA

2. Secondary Outcome: The Distribution of Changes From Baseline in the Prescribed ESA Dose Between the Two Treatment Arms
Description: The change from baseline in prescribed ESA dose at end-of-treatment was categorized as being greater than or equal to 25%, 10 to less than 25%, -10 to 10%, greater than -25 to -10% and less than or equal to -25%. The number of subjects in each treatment group that fit each category was compared.
Time Frame: ESA dose is monitored and recorded at each dialysis session for 36 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | SFP in Liquid Bicarbonate | Placebo: Conventional Liquid Bicarbonate
Number analyzed (Participants) | 52 | 51
Participants
  ESA dose change > or = to 25% | 16 | 20
  ESA dose change >10 to 25% | 5 | 4
  ESA dose change > -10% to 10% | 12 | 9
  ESA dose change > -25% to -10% | 3 | 3
  ESA dose change < or = to -25% | 16 | 15
Statistical Analysis 1: Comparison: SFP in Liquid Bicarbonate vs Placebo: Conventional Liquid Bicarbonate; Test type: Superiority or Other; p = 0.915, Cochran-Mantel-Haenszel

3. Secondary Outcome: Stability of Hemoglobin Over Time (Maintenance of Hemoglobin Between 9.5-11.5 g/dL.
Description: The number of patients in each treatment group who had maintained their hemoglobin between 95 and 115 grams/liter at the end of treatment was quantified.
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SFP in Liquid Bicarbonate | Placebo: Conventional Liquid Bicarbonate
Number analyzed (Participants) | 52 | 51
Participants | 30 | 30
Statistical Analysis 1: Comparison: SFP in Liquid Bicarbonate vs Placebo: Conventional Liquid Bicarbonate; Test type: Superiority or Other; p = 0.6714, Cochran-Mantel-Haenszel

4. Secondary Outcome: The Amount of Supplemental Intravenous (IV) Iron Needed During Study Participation.
Description: The absolute amount of IV iron administered to subjects in each treatment group was divided by the number of weeks on study and the number of subjects per treatment group such that the mean dose of IV iron (mg) per week per subject (for the entire treatment group) was calculated.
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: mg per week per subject
Arm/Group | SFP in Liquid Bicarbonate | Placebo: Conventional Liquid Bicarbonate
Number analyzed (Participants) | 52 | 51
mg per week per subject | 23.5 (54.22) | 45.6 (62.78)
Statistical Analysis 1: Comparison: SFP in Liquid Bicarbonate vs Placebo: Conventional Liquid Bicarbonate; Test type: Superiority or Other; p = 0.028, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Comparison of Iron Delivery to the Erythron From Baseline to End of Treatment Between the Treatment Groups.
Description: Iron delivery to the erythron was estimated by Hgb generation in response to erythropoietin (ERI, calculated as ESA dose/Hgb). In addition, ERI was also divided by body weight in kilograms to obtain a modified ERI (ERI/kg).
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: Units/kilogram/week/gram/liter
Arm/Group | SFP in Liquid Bicarbonate | Placebo: Conventional Liquid Bicarbonate
Number analyzed (Participants) | 52 | 51
Units/kilogram/week/gram/liter
  baseline | 10.43 (6.457) | 10.38 (6.471)
  end of treatment | 11.71 (9.808) | 14.67 (13.804)
Statistical Analysis 1: Comparison: SFP in Liquid Bicarbonate vs Placebo: Conventional Liquid Bicarbonate; Test type: Superiority or Other; p = 0.361, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: Safety Population: Subjects who received any amount of study drug, including those who receive the wrong treatment.
Arm/Group | SFP in Liquid Bicarbonate | Placebo: Conventional Liquid Bicarbonate
Serious Adverse Events (participants affected / at risk) | 18/54 | 20/49
Other Adverse Events (participants affected / at risk) | 50/54 | 46/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SFP in Liquid Bicarbonate (N=54) | Placebo: Conventional Liquid Bicarbonate (N=49)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 (3) | 2 (2)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 2 (2)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 2 (3)
SUDDEN CARDIAC DEATH (General disorders) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 2 (2)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 2 (2)
DIABETIC FOOT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0)
GANGRENE (Infections and infestations) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GASTROINTESTINAL ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 1 (1)
VASCULAR DEMENTIA (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 2 (2)
BRAIN STEM HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 1 (1)
AZOTAEMIA (Renal and urinary disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DIABETIC NEUROPATHIC ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 2 (2) | 0 (0)
MALIGNANT HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SFP in Liquid Bicarbonate (N=54) | Placebo: Conventional Liquid Bicarbonate (N=49)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 18 (145) | 20 (184)
HAEMODIALYSIS-INDUCED SYMPTOM (Injury, poisoning and procedural complications) | 12 (19) | 6 (13)
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 10 (14) | 8 (17)
NAUSEA (Gastrointestinal disorders) | 8 (12) | 7 (11)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 8 (9) | 6 (6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (11)
HEADACHE (Nervous system disorders) | 7 (16) | 8 (16)
ASTHENIA (General disorders) | 7 (11) | 3 (3)
BRADYCARDIA (Cardiac disorders) | 7 (15) | 2 (3)
VOMITING (Gastrointestinal disorders) | 6 (7) | 8 (10)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (8) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (6) | 4 (4)
CONSTIPATION (Gastrointestinal disorders) | 5 (5) | 1 (1)
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 4 (7) | 10 (17)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (10)
DIZZINESS (Nervous system disorders) | 4 (9) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (8) | 4 (7)
ANXIETY (Psychiatric disorders) | 4 (4) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
HYPERTENSION (Vascular disorders) | 4 (5) | 2 (2)
PNEUMONIA (Infections and infestations) | 4 (4) | 2 (2)
VASCULAR GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 4 (5) | 1 (8)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 (12) | 5 (15)
PYREXIA (General disorders) | 3 (4) | 5 (5)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 (4) | 3 (3)
EXCORIATION (Injury, poisoning and procedural complications) | 3 (3) | 3 (4)
METABOLIC ALKALOSIS (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
ANAEMIA (Blood and lymphatic system disorders) | 3 (5) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 3 (4) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 2 (2) | 4 (7)
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 2 (5) | 4 (4)
ANGINA PECTORIS (Cardiac disorders) | 2 (3) | 3 (9)
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 2 (3) | 3 (5)
FALL (Injury, poisoning and procedural complications) | 2 (3) | 3 (8)
LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 3 (5)
INSOMNIA (Psychiatric disorders) | 1 (1) | 3 (3)
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 (0) | 3 (3)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 (0) | 3 (3)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No study results may be submitted for publication without Sponsor's prior written consent. Within 60 days from submission to Sponsor's review, Sponsor may withhold the consent. 1st publication of results is made in conjunction with the presentation of a joint, multicenter publication of results with certain PIs from all sites contributing data.